CLINICAL TRIAL: NCT04572360
Title: Would Cardiorespiratory Exercise and Chinese Herbal Medicine Facilitate Rehabilitation Among Post-discharge Patients With COVID-19? Clinical Efficacy and Mechanisms
Brief Title: Cardiorespiratory Exercise & Chinese Medicine for Rehabilitation of Discharged Coronavirus Disease (COVID-19) Patients
Acronym: Covid19Reh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other); The Hong Kong Polytechnic University (Other); University of South Wales (Other); Yale University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKCOVID19Rehab
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: COVID-19; Cardiorespiratory Exercise; Chinese Medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A triple-blinded, randomized, parallel groups, controlled clinical trial. A total of 172 eligible patients will be randomized 1:1:1:1 into four groups: cardiorespiratory exercise plus Chinese herbal medicines group, cardiorespiratory exercise group, Chinese herbal medicines group and waiting list group for 12-week (3 months) with 12-week follow-up period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patients and investigators will be blinded to the assigned groups. Patients will be allocated at a ratio of 1:1:1:1, the randomization will be carried out by Statistical Analysis System 9.3 (SAS 9.3) statistical software. (Descript how the blinding works here) One copy of the blind codes will be held by the project responsible unit. The statistician will be blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cardiorespiratory Exercise plus Chinese Herbal Medicines Group (Experimental): Includes:
  1.12-week progressive & individualized exercise, 60mins/session, 3 sessions/week, total 36 exercise sessions. Components: a set of home-based tele-exercise sessions with remote monitoring of vital signs; individualized action plan to perform various daily physical activities; educational sessions on self-management & habit formation; access to a call center; & counselling sessions to enhance motivation to regularly engage in daily physical activities.
  2.Chinese herbal formula of Modified Bai He Gu Jin Tang prescribed in granules, 10g/day (5g dissolved in 200ml of hot water, b.i.d), twice/day after breakfast & dinner, 7days/week for 12 weeks.
  Interventions: Other: Cardiorespiratory Exercise; Other: Modified Bai He Gu Jin Tang
- Cardiorespiratory Exercise Group (Experimental): Includes:
  A 12-week progressive & individualized exercise, 60mins/session, 3 sessions/week, total 36 exercise sessions. Components: a set of home-based tele-exercise sessions with remote monitoring of vital signs; individualized action plan to perform various daily physical activities; educational sessions on self-management & habit formation; access to a call center; & counselling sessions to enhance motivation to regularly engage in daily physical activities.
  Interventions: Other: Cardiorespiratory Exercise
- Chinese Herbal Medicines Group (Experimental): Includes:
  Chinese herbal formula of Modified Bai He Gu Jin Tang prescribed in granules, 10g/day (5g dissolved in 200ml of hot water, b.i.d), twice/day after breakfast & dinner, 7days/week for 12 weeks.
  Interventions: Other: Modified Bai He Gu Jin Tang
- Waiting List Group (No Intervention): The waiting list control sign will be adopted to conceal allocation results from the patients and further to reduce selection and confounding bias and increase their adherence to the study. Patients in the waiting list control group will receive no treatment in the study period (including a 12-week intervention period and a 12-week follow-up period). However, they will receive Chinese herbal medicines after the completion of the study (i.e., after the 3rd wave of measurements in the 25th weeks).

INTERVENTIONS:
Other: Cardiorespiratory Exercise — Each exercise session (40-60 minutes) will include warm-up, aerobic training, resistance training, cool-down, as well as inspiratory muscle training
  Arms: Cardiorespiratory Exercise Group; Cardiorespiratory Exercise plus Chinese Herbal Medicines Group
Other: Modified Bai He Gu Jin Tang — The Chinese herbal formula of Modified Bai He Gu Jin Tang will be prescribed in granules. A dose of 10g a day (5g, b.i.d) will be ingested. Patients will dissolve a sachet of granules (5.0g) in 200ml of hot water, twice a day after breakfast and dinner, seven days a week for three months.
  Arms: Cardiorespiratory Exercise plus Chinese Herbal Medicines Group; Chinese Herbal Medicines Group

SUMMARY:
Rehabilitation interventions can help to address the consequences of COVID-19, which include medical, physical, cognitive, and psychological related problems. The specific aims of this project are to investigate the effects of a 12-week exercise program on pulmonary fibrosis in recovering COVID-19 patients. A further aim will be to examine how Chinese herbal medicines, gut microbiome, and metabolites regulate immune function and possibly autoimmune deficiency in the rehabilitation process.

DETAILED DESCRIPTION:
The study will develop a new paradigm for patient rehabilitation needed now and in the future. The specific aims of this project are to investigate the effects of a 12-week program with cardiorespiratory exercise and Chinese herbal medicine on recovering COVID-19 patients and to collect qualitative and quantitative data to examine loneliness, anxiety, depression, quality of life, and mental health. A further aim will be to examine how Chinese herbal medicines, gut microbiome, and the metabolites regulate immune function, intestinal permeability, and possibly autoimmune deficiency (AID) in the pathological recovery/rehabilitation process.

In this multicenter, triple-blinded, randomized, parallel groups, controlled clinical trial, the investigator will recruit adult patients with COVID-19 and have been discharged from the hospital in Hong Kong and the Chinese Mainland.

A total of 172 eligible patients will be randomized 1:1:1:1 into four groups: cardiorespiratory exercise plus Chinese herbal medicines group, cardiorespiratory exercise group, Chinese herbal medicines group, and waiting list group for 12-week (3 months) with 12-week follow-up period.

A 4-week pilot study will be conducted to test patient recruitment and maintenance, data collection, instrumentation, and observing the adaptability and practicality of the intervention. Amendments will be made if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and above;
2. a percentage of predicted forced vital capacity (FVC) <90%, and/or a percentage of predicted carbon monoxide diffusing capacity < 90% (King 2014);
3. able to communicate in Cantonese.

Exclusion Criteria:

1. having acute exacerbations in the 12-week preceding recruitment patients;
2. having any contraindications for exercise (e.g., physical disability, uncontrolled mental disorders, unstable heart disease, unable to perform muscle strength tests)
3. Female - Pregnant or plan to become pregnant in the next 1 year
4. Unable to communicate in Cantonese or Mandarin
5. Currently participating in other similar rehabilitation programs or research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) in Cardiorespiratory Fitness Test | 6 months
  To assess the functional exercise capacity that reflects daily physical activities and to measure the distance the participant is able to walk over six minutes on a hard, flat surface.
  Items measured during 6MWT are:
  * Distance Walked (m)
  * Number of Rests
Blood Pressure | 6 months
  Blood pressure (Systolic/Diastolic) in mmHg will be measured before & after 6MWT
Heart Rate | 6 months
  Heart rate in beats per minute will be measured before & after 6MWT
Peripheral oxygen saturation (SpO2) | 6 months
  SpO2 in % will be measured before & after 6MWT
Borg Dyspnea Scale | 6 months
  The Borg Category Ratio 10 (CR10) Scale® (Borg Dyspnea Scale), will be used to rate the patients' dyspnea and overall fatigue level. At the beginning and end the end of the 6 MWT. The scale will also be used during Cardiopulmonary Exercise Test (CPET).
  Scale:
  0=Rest; 0.5=Really Really Easy; 1=Really Easy; 2=Easy; 3=Moderate; 4=Sort of Hard; 5,6=Hard; 7,8,9=Really Hard; 10=Maximal
Body composition - Segmental Muscle Mass | 6 months
  Bio-impedance analysis approach will be used to assess patient's segmental muscle mass in percentage (%).
Body composition - Body Mass Index (BMI) | 6 months
  A stadiometer will be used to measure stature (in metres) and weight is measured in kg to calculate body mass index (BMI) .
  Body Mass Index (BMI): weight (in kilograms) divided by the square of your height (in metres)
Body composition - Anatomical Circumferences | 6 months
  Anatomical circumferences - waist (cm) & Hip (cm) will be measured using a steel measuring tape, to calculate the Waist-to-Hip Ratio.
FVC (L) in Lung function Test using Spirometry | 6 months
  Forced vital capacity test (FVC) will be measured and used to calculate FEV1/FVC ratio to assess the functional severity and capacity of the patient's lung.
FEV1 (L) in Lung function Test using Spirometry | 6 months
  Forced expiratory volume (FEV1) will be measured and used to calculate FEV1 /FVC ratio to assess the functional severity and capacity of the patient's lung.
MVV (L/min) in Lung function Test using Spirometry | 6 months
  Maximal Voluntary Ventilation (MVV) measures peak performance of the lungs and respiratory muscles to assess overall pulmonary ventilation.
Fractional exhaled Nitric Oxide (FeNO) | 6 months
  Fractional exhaled Nitric Oxide (FeNO), the results will be in parts per billion (ppb) of nitric oxide in patient's breath, will be used to assess inflammatory response to exercise and medicinal intervention.
Diffusing capacity of the lungs for carbon monoxide (DLCO) | 6 months
  Diffusing capacity of the lungs for carbon monoxide (DLCO), measured in millilitre/minute/Kilopascal (ml/min/kPa), will be used to evaluate gas diffusion in the lungs.
Cardiopulmonary Exercise Test (CPET) - Work Rate(WR) | 6 months
  CPET provides information concerning the level of exercise that the patient can perform without undue stress. The test results will guide the research team regarding exercise prescription for physical rehabilitation methodologies, and provides quantitative evidence of the benefits of a rehabilitation program as well as information on the mechanism(s) involved.
  Work Rate(WR), an incremental ergometry exercise test, will be used to assess the cellular, cardiovascular, and ventilatory systems' responses under precise conditions of metabolic stress
Cardiopulmonary Exercise Test (CPET) - Breath by Breath Measurements of Minute ventilation (VE) | 6 months
  Breath by breath measurements of minute ventilation (VE) in L/min will be measured and used to calculate ventilatory efficiency - VE/VCO2 and VE/VO2, ventilatory equivalents for carbon dioxide and oxygen.
Cardiopulmonary Exercise Test (CPET) - CO2 output (VCO2) | 6 months
  CO2 output (VCO2) in L/min, will be measured and used to calculate ventilatory efficiency - VE/VCO2, ventilatory equivalents for carbon dioxide.
Cardiopulmonary Exercise Test (CPET) - O2 uptake (VO2) | 6 months
  O2 uptake (VO2) in L/min, will be measured and used to calculate ventilatory efficiency - VE/VO2, ventilatory equivalents for oxygen.
Change in Chinese Medicine (CM) Diagnostic Pattern & Clinical Characteristics using CM Syndrome Differentiation Assessment | Change from baseline the CM Diagnostic Pattern & Clinical Characteristics at 6 months
  The changes in participants' health as characterized by CM diagnostic pattern & clinical characteristics using CM Syndrome Differentiation according to the Guidelines for Chinese Medicine New Drug Clinical Study (China Medical Science Press, 2002) will be assessed.
Change in Body Constitution Scores using Body Constitution Questionnaires Assessment | Change from baseline the Body Constitution at 6 months
  The changes in participants' health as characterized by body constitution scores using the Body Constitution Questionnaires for the nine specific types of body constitutions will be assessed on each visit during the treatment and follow up period.

SECONDARY OUTCOMES:
Blood Biochemistry Tests - Serum Levels of Insulin (pmol/l) | 6 months
  Venous blood will be drawn & after coagulation at room temperature for 30 minutes, the samples will be centrifuged at 3000 rpm for 20 minutes. Serum as supernatant will be extracted & stored at -80˚C until assay. Serum levels of insulin will be assessed by a commercially available Enzyme-linked immunosorbent Assay (ELISA) kit (Merck).
Blood Biochemistry Tests - Prothrombin Time (seconds) | 6 months
  The Prothrombin time test will be used to measure blood coagulation. Venous blood will be collected by venepuncture in a tube with sodium citrate. Plasma will be isolated after centrifugation at 1000rpm for 30 min, 4°C. Thromboplastin will be added into the plasma and kept at 37°C for two minutes. Calcium chloride will be added to the mixture, and the plasma is allowed to coagulate. The time needed for the coagulation will be recorded as the Prothrombin Time.
Quality of Life - Personal Wellbeing Index - Chinese Version (Adult) | 6 months
  Quality of life (QoL) will be measured using the Personal Well-being Index-Chinese Version (PWI-C). It is a subjective QoL measure with questionnaires that have been translated and validated.
  Questions included are:
  How satisfied are you with…?"
  1. your standard of living ?
  2. your health ?
  3. what you are achieving in life ?
  4. your personal relationships ?
  5. how safe you feel ?
  6. feeling part of your community ?
  7. your future security ?
  Answers are measured using scale from zero to 10 (0...1…2...3...4…5...6...7...8...9…10).
  Zero means feel no satisfaction at all; 10 means feel completely satisfied.
Other mental health-related measures - Depression Anxiety Stress Scale (DASS-21) | 6 months
  Anxiety and stress will be measured using the Chinese version of the Depression Anxiety Stress Scale (DASS-21). The scale will discriminate between the negative emotional syndromes of depression, anxiety, and stress in Chinese populations. Only the subscales of anxiety and stress will be used.
  The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic nonspecific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive & impatient.
  The rating scale is as follows:
  0=Did not apply to me at all
  1. Applied to me to some degree, or some of the time
  2. Applied to me to a considerable degree or a good part of time
  3. Applied to me very much or most of the time
  Scores are calculated by summing the scores for the relevant items. Higher scores indicate greater degrees of anxiety and stress.
Other mental health-related measures - Revised UCLA Loneliness Scale (R-UCLA) | 6 months
  Loneliness will be measured using the Revised UCLA Loneliness Scale (R-UCLA). It consists of 20 items and participants are to indicate how often they feel the way described by placing a check in the space provided, using the following scale:
  1. Never
  2. Rarely
  3. Sometimes
  4. Often
  Score scale for item 1,5,6,9,10,15,16,19,20 are reversed, and score for each item then summed together. Higher scores indicate greater degrees of loneliness.
Other mental health-related measures - General Health Questionnaire (GHQ) | 6 months
  General mental health will be measured using the General Health Questionnaire (GHQ), which is commonly used to screen minor psychiatric symptoms (Hu 2007).
  It consists of 12 items, beginning by asking "Have you recently…", each assessing the severity of a mental problem over the past few weeks using a 4-point scale of: (always) 0...1…2…3 (never).
  The score was used to generate a total score ranging from 0 to 36, with higher scores indicating worse conditions.
Gut microbiome Test | 6 months
  Patient is to self-sample morning first feces & immediately freeze it in a home freezer (-20℃) & transport to facilities in a provided freezer pack stored at -80℃. Total DNA of 200 mg fecal samples will be extracted & purified. The DNA concentration & size distribution will be estimated by a Nano drop instrument & agarose gel electrophoresis respectively. The DNA one paired-end (PE) library will be prepared using a DNA high-throughput (HT) Sample Prep Kit, & whole-genome shotgun sequencing of samples will be carried out by the Illumina platform. The high quality sequences will be mapped with the published gene catalog of reference genes in the human gut microbiome (Li 2014). Taxonomic assignment of the predicted genes and Kyoto Encyclopedia of Genes & Genomes (KEGG) analysis will be performed as described (Feng 2015). Relative abundances of phyla, genera, species, & Kegg Orthology (KOs) will be calculated from the relative abundances of the respective genes.
Metabolomics-related Measurement of Depression - Metabolomics Analysis | 6 months
  Metabolomics analysis of selected neurotransmitters as potential markers of depression: Ultra-performance liquid chromatography triple quadrupole mass spectrometry will be used to quantitatively measure the metabolites selected (neurotransmitters) as potential markers of depression. Briefly, an aliquot of 40 μl of urine or plasma will be spiked with 10 μL of internal standard (L-4-chlorophenylalanine in water, 30 μg/mL), and extracted with 200 μL of acetonitrile and methanol (9:1, v/v). The mixture will be vortexed and centrifuged. After centrifugation, the supernatant will be transferred to the sampling vials and subject to analysis. The raw data generated will be processed using the Target Lynx Applications Manager Version 4.1 (Waters Corp., Milford, MA) for targeted metabolite annotation and to obtain calibration equations and the concentration of each metabolite in the samples Metabolomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Julien Baker, Ph.D, D.Sc, Study Chair — Department of Sport, Physical Education and Health, Hong Kong Baptist University
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be deidentified and available for anyone who wish to access the data immediately following publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after the completion of study.
Access Criteria: All researchers can get the information by sending requests to the study contact person.

REFERENCES:
- [Derived] Gao Y, Zhong LLD, Quach B, Davies B, Ash GI, Lin ZX, Feng Y, Lau BWM, Wagner PD, Yang X, Guo Y, Jia W, Bian Z, Baker JS. COVID-19 Rehabilitation With Herbal Medicine and Cardiorespiratory Exercise: Protocol for a Clinical Study. JMIR Res Protoc. 2021 May 26;10(5):e25556. doi: 10.2196/25556. PMID 33970864